CLINICAL TRIAL: NCT02538783
Title: A Randomized Trial of Financial Incentives for Maintenance of Weight Loss
Brief Title: The Weigh Forward, Financial Incentives for Maintenance of Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Duke University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 823005; 1R01AG045045-01 (NIH)
Record Dates: First submitted 2015-08-31; First posted 2015-09-02 (Estimated); Results first posted 2019-01-14 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2018-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Participants will receive weekly tips and weekly feedback for months 1-6 and will be observed without intervention in Phase II (months 7-12). The weekly feedback will pertain to whether or not the participant met his/her goal of weighing at least 6/7 days. The weekly tips will give information and suggestions on how to make it easier to weigh-in most days of the week. No financial incentive other than for the midpoint and end of study surveys will be given.
- Escalating lottery (Experimental): Participants will receive weekly tips and weekly feedback for months 1-6 and will be observed without intervention in Phase II (months 7-12). The weekly feedback will pertain to whether or not the participant met his/her goal of weighing at least 6/7 days. The weekly tips will give information and suggestions on how to make it easier to weigh-in most days of the week. In addition to the incentives for midpoint and end of study surveys, participants who meet their weekly goal (weighing in 6 of 7 days) will be eligible for the weekly lottery during the first 6 months of the study. The expected weekly winning for the lottery is $3.55 in week 1 and this expected value will increase by $0.43 per week for each week the participant achieves their goal of weighing 6/7 days. All incentive earnings will be paid out on a monthly basis.
  Interventions: Behavioral: Escalating Lottery

INTERVENTIONS:
Behavioral: Escalating Lottery — Participants in the lottery arms will receive financial incentives as part of the intervention. See arm descriptions for more detail.
  Arms: Escalating lottery

SUMMARY:
This study aims to evaluate the effectiveness of financial incentives in improving and maintaining weight loss.

DETAILED DESCRIPTION:
The study will evaluate the effectiveness of financial incentives in improving maintenance of weight loss. The investigators propose a 2-arm randomized controlled trial in which 258 participants who lose at least 5 kgs in a weight loss program will be randomized to one of the following: 1) daily weigh-ins and weekly feedback, 2) daily weigh-ins,weekly feedback, and a weekly escalating lottery-based financial incentive.

Study participants will be obese volunteers recruited from a major community-based weight loss program (Weight Watchers), who have lost at least 5kg during the 4-6 months prior to enrolling in the study. Upon enrollment, these participants will have an active online membership with Weight Watchers. Among these participants, the following will be assessed: 1. Assess the effectiveness of escalating lottery rewards, relative to the control group, on maintenance of weight loss over the ensuing 6 months (Phase I); 2.The degree to which weight loss is maintained in the intervention group relative to usual care during the 6 months following the cessation of the interventions (Phase II).

During Phase I, incentives will be provided to some study participants (escalating lottery arm) for the first 6 months and participants will be followed for 6 more months to examine effects following cessation of incentives.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 30-80
* BMI between 30 and 45 prior to starting Weight Watchers
* Have a documented weight loss of at least 5kg in the past 4-6 months before enrolling
* Stable health
* Have an online Weight Watchers membership

Exclusion Criteria:

* Substance abuse
* Bulimia nervosa or related behaviors
* Pregnancy or breast feeding
* Medical contraindications to counseling about diet, physical activity, or weight reduction
* Unstable mental illness
* Screen positive for pathological gambling on the basis of the 10 item DSM-IV criteria (excluded if meets 5 or more criteria)
* Individuals unable to read consent forms or fill out surveys in English

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2016-05-01; Primary Completion 2017-11-13 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Clinical Guidelines on the Identification, Evaluation, and Treatment of Overweight and Obesity in Adults--The Evidence Report. National Institutes of Health. Obes Res. 1998 Sep;6 Suppl 2:51S-209S. No abstract available. PMID 9813653
- [Background] Office of the Surgeon General (US); Office of Disease Prevention and Health Promotion (US); Centers for Disease Control and Prevention (US); National Institutes of Health (US). The Surgeon General's Call To Action To Prevent and Decrease Overweight and Obesity. Rockville (MD): Office of the Surgeon General (US); 2001. Available from http://www.ncbi.nlm.nih.gov/books/NBK44206/ PMID 20669513
- [Background] Flegal KM, Carroll MD, Ogden CL, Johnson CL. Prevalence and trends in obesity among US adults, 1999-2000. JAMA. 2002 Oct 9;288(14):1723-7. doi: 10.1001/jama.288.14.1723. PMID 12365955
- [Background] Ogden CL, Carroll MD, Curtin LR, McDowell MA, Tabak CJ, Flegal KM. Prevalence of overweight and obesity in the United States, 1999-2004. JAMA. 2006 Apr 5;295(13):1549-55. doi: 10.1001/jama.295.13.1549. PMID 16595758
- [Background] Adams KF, Schatzkin A, Harris TB, Kipnis V, Mouw T, Ballard-Barbash R, Hollenbeck A, Leitzmann MF. Overweight, obesity, and mortality in a large prospective cohort of persons 50 to 71 years old. N Engl J Med. 2006 Aug 24;355(8):763-78. doi: 10.1056/NEJMoa055643. Epub 2006 Aug 22. PMID 16926275
- [Background] Daviglus ML, Liu K, Yan LL, Pirzada A, Manheim L, Manning W, Garside DB, Wang R, Dyer AR, Greenland P, Stamler J. Relation of body mass index in young adulthood and middle age to Medicare expenditures in older age. JAMA. 2004 Dec 8;292(22):2743-9. doi: 10.1001/jama.292.22.2743. PMID 15585734
- [Background] Finkelstein EA, Trogdon JG, Brown DS, Allaire BT, Dellea PS, Kamal-Bahl SJ. The lifetime medical cost burden of overweight and obesity: implications for obesity prevention. Obesity (Silver Spring). 2008 Aug;16(8):1843-8. doi: 10.1038/oby.2008.290. Epub 2008 May 29. PMID 18535543
- [Background] Nordmann AJ, Nordmann A, Briel M, Keller U, Yancy WS Jr, Brehm BJ, Bucher HC. Effects of low-carbohydrate vs low-fat diets on weight loss and cardiovascular risk factors: a meta-analysis of randomized controlled trials. Arch Intern Med. 2006 Feb 13;166(3):285-93. doi: 10.1001/archinte.166.3.285. PMID 16476868
- [Background] Gardner CD, Kiazand A, Alhassan S, Kim S, Stafford RS, Balise RR, Kraemer HC, King AC. Comparison of the Atkins, Zone, Ornish, and LEARN diets for change in weight and related risk factors among overweight premenopausal women: the A TO Z Weight Loss Study: a randomized trial. JAMA. 2007 Mar 7;297(9):969-77. doi: 10.1001/jama.297.9.969. PMID 17341711
- [Background] Methods for voluntary weight loss and control. NIH Technology Assessment Conference Panel. Consensus Development Conference, 30 March to 1 April 1992. Ann Intern Med. 1993 Oct 1;119(7 Pt 2):764-70. PMID 8363212
- [Background] Giuffrida A, Torgerson DJ. Should we pay the patient? Review of financial incentives to enhance patient compliance. BMJ. 1997 Sep 20;315(7110):703-7. doi: 10.1136/bmj.315.7110.703. PMID 9314754
- [Background] Kane RL, Johnson PE, Town RJ, Butler M. A structured review of the effect of economic incentives on consumers' preventive behavior. Am J Prev Med. 2004 Nov;27(4):327-52. doi: 10.1016/j.amepre.2004.07.002. PMID 15488364
- [Background] Volpp KG, Gurmankin Levy A, Asch DA, Berlin JA, Murphy JJ, Gomez A, Sox H, Zhu J, Lerman C. A randomized controlled trial of financial incentives for smoking cessation. Cancer Epidemiol Biomarkers Prev. 2006 Jan;15(1):12-8. doi: 10.1158/1055-9965.EPI-05-0314. PMID 16434580
- [Background] Volpp KG, Troxel AB, Pauly MV, Glick HA, Puig A, Asch DA, Galvin R, Zhu J, Wan F, DeGuzman J, Corbett E, Weiner J, Audrain-McGovern J. A randomized, controlled trial of financial incentives for smoking cessation. N Engl J Med. 2009 Feb 12;360(7):699-709. doi: 10.1056/NEJMsa0806819. PMID 19213683
- [Background] Volpp KG, John LK, Troxel AB, Norton L, Fassbender J, Loewenstein G. Financial incentive-based approaches for weight loss: a randomized trial. JAMA. 2008 Dec 10;300(22):2631-7. doi: 10.1001/jama.2008.804. PMID 19066383
- [Background] Flegal KM, Graubard BI, Williamson DF, Gail MH. Excess deaths associated with underweight, overweight, and obesity. JAMA. 2005 Apr 20;293(15):1861-7. doi: 10.1001/jama.293.15.1861. PMID 15840860
- [Background] Must A, Spadano J, Coakley EH, Field AE, Colditz G, Dietz WH. The disease burden associated with overweight and obesity. JAMA. 1999 Oct 27;282(16):1523-9. doi: 10.1001/jama.282.16.1523. PMID 10546691
- [Background] The sixth report of the Joint National Committee on prevention, detection, evaluation, and treatment of high blood pressure. Arch Intern Med. 1997 Nov 24;157(21):2413-46. doi: 10.1001/archinte.157.21.2413. PMID 9385294
- [Background] Eckel RH. Obesity and heart disease: a statement for healthcare professionals from the Nutrition Committee, American Heart Association. Circulation. 1997 Nov 4;96(9):3248-50. doi: 10.1161/01.cir.96.9.3248. No abstract available. PMID 9386201

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Escalating Lottery
Started | 130 | 129
Completed | 130 | 128
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Escalating Lottery | Total
Number analyzed (Participants) | 130 | 128 | 258
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 122 | 124 | 246
  >=65 years | 8 | 4 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.2 (10.6) | 46.9 (10.2) | 48 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 112 | 225
  Male | 17 | 16 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 6 | 15
  Not Hispanic or Latino | 121 | 122 | 243
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 8 | 12
  White | 120 | 115 | 235
  More than one race | 4 | 1 | 5
  Unknown or Not Reported | 1 | 2 | 3
Education [Count of Participants; unit: Participants]
  High School or less | 22 | 11 | 33
  Some college | 42 | 34 | 76
  College degree | 33 | 41 | 74
  Post graduate | 33 | 42 | 75
Income [Count of Participants; unit: Participants]
  <$50,000 | 15 | 14 | 29
  $50,000 to $99,000 | 62 | 65 | 127
  $100,000 to $149,000 | 41 | 35 | 76
  >=$150,000 | 12 | 14 | 26
Household Size [Mean (Standard Deviation); unit: people per household] | 2.8 (1.3) | 3.2 (1.6) | 3 (1.4)
BMI at randomization [Mean (Standard Deviation); unit: kg/m^2] | 31.7 (3.7) | 32.6 (4.2) | 32.1 (3.9)
Weight loss prior to randomization [Mean (Standard Deviation); unit: kilograms] | 11.5 (4.3) | 11.8 (4.1) | 11.6 (4.2)
Willing to give up something today in order to benefit in the future [Count of Participants; unit: Participants] — The score is measured by the respondent's answer to this question: How do you see yourself? Are you a person who is generally willing to give up something today in order to benefit from that in the future, or are you not willing to do so? Please use a scale from 1 to 10, where 1 means you are "completely unwilling to give up something today" and 10 means you are "very willing to give up something today". Selecting 0-3 on the scale means the participant is most adverse to risks, 4-7 indicates moderate adverse to risks, and 8-10 is least averse to risks.
  Participants
    Most averse to risks | 44 | 45 | 89
    Moderate averse to risks | 70 | 65 | 135
    Least averse to risks | 16 | 18 | 34
Postpone things even though it would be better to get done right away [Count of Participants; unit: Participants] — The Procrastinator Score is measured by the respondent's answer to the question: How well does the following statement describe you as a person? I tend to postpone things even though it would be better to get them done right away. Use a scale from 0 to 10, where 0 means "does not describe me at all" and a 10 means "describes me perfectly". Selecting 0-3 on the scale means the participant is most adverse to risks, 4-7 indicates moderate adverse to risks, and 8-10 is least averse to risks.
  Participants
    Most averse to risks | 44 | 45 | 89
    Moderate averse to risks | 70 | 65 | 135
    Least averse to risks | 16 | 18 | 34
Baseline IPAQ Level [Count of Participants; unit: Participants] — Physical activity categories:
  Scoring a HIGH level on the IPAQ means physical activity levels equate to approximately one hour of activity per day or more at least a moderate intensity activity level.
  Scoring a MODERATE level of physical activity on the IPAQ means you are doing some activity more than likely equivalent to half an hour of at least moderate intensity physical activity on most days.
  Scoring a LOW level of physical activity on the IPAQ means that you are not meeting any of the criteria for either MODERATE of HIGH levels of physical activity
  Participants
    Low | 20 | 28 | 48
    Moderate | 52 | 55 | 107
    High | 58 | 44 | 102
    Missing | 0 | 1 | 1
Baseline MVPA minutes/week [Median (Inter-Quartile Range); unit: Minutes per week] | 180 [30 to 390] | 145 [50 to 270] | 150 [40 to 305]
Baseline Walking minutes/week [Median (Inter-Quartile Range); unit: Minutes per week] | 210 [100 to 480] | 210 [105 to 420] | 210 [100 to 420]
Eating behaviors by Three Factor Questionnaire [Mean (Standard Deviation); unit: scores on a scale] — The TFEQ consists of 18 items on a 4-point response scale (definitely true/mostly true/mostly false/definitely false). Responses to each of the 18 items are given a score between 1 and 4 and item scores are summated into scale scores for cognitive restraint, uncontrolled eating, and emotional eating. The raw eating scale scores are transformed to a 0-100 scale [((raw score - lowest possible raw score)/possible raw score range) × 100] Higher scores in the respective scales are indicative of greater cognitive restraint, uncontrolled, or emotional eating
  scores on a scale
    Baseline cognitive restraint | 63.2 (12.9) | 64.1 (15.6) | 63.7 (14.3)
    Baseline uncontrolled eating | 41.8 (17.9) | 42.7 (17.9) | 42.2 (17.9)
    Baseline emotional eating | 51.4 (25.4) | 53.9 (24.5) | 52.6 (24.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight, Baseline and 6 Months
Description: Among participants who lost 5 kg or more of baseline weight prior to randomization, assess the effectiveness of escalating lottery rewards, relative to the control group, on maintenance of weight loss after 6 months of intervention
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Control | Escalating Lottery
Number analyzed (Participants) | 130 | 128
Kilograms | -1.9 (5.9) | -1.1 (5.7)

2. Primary Outcome: Change in Weight, 6 Months and 12 Months
Description: Among participants who lost 5 kg or more of baseline weight prior to randomization, assess the degree to which weight loss is maintained in the intervention groups relative to usual care during the 6 months following the cessation of the interventions
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Control | Escalating Lottery
Number analyzed (Participants) | 130 | 128
Kilograms | -0.6 (8.2) | 0.2 (8.1)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 1 year (length of time in study).
Arm/Group | Control | Escalating Lottery
All-Cause Mortality (participants affected / at risk) | 0/130 | 0/128
Serious Adverse Events (participants affected / at risk) | 5/130 | 3/129
Other Adverse Events (participants affected / at risk) | 4/130 | 2/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=130) | Escalating Lottery (N=129)
Diagnosis of multiple sclerosis (Immune system disorders) | 1 (1) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Soft tissue sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Ankle infection (Infections and infestations) | 1 (1) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Full right hip replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=130) | Escalating Lottery (N=129)
Knee injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Outpatient foot surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Outpatient knee surgery (Surgical and medical procedures) | 2 (2) | 0 (0)
Outpatient hernia surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Outpatient bladder and rectum repair surgery (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/83/NCT02538783/Prot_SAP_000.pdf